CLINICAL TRIAL: NCT01393275
Title: Effects of Exercise Intervention in Patients With Type 2 Diabetes - Strength Endurance Exercise Intervention Versus Combination of Strength Endurance Exercise Intervention and Rehabilitation Exercise Intervention
Brief Title: Effects of Exercise Intervention and Rehabilitation Exercise Intervention in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Sportpark Zwickau, Germany (Unknown); Sportpark Glauchau, Germany (Unknown); Comenius University (Other)
Responsible Party: Principal Investigator, Andree Hillebrecht, Akad. Rat, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gi-01-2010
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Diabetes; Diabetes Mellitus, Non-Insulin-Dependent
Keywords: diabetes; exercise; intervention; rehabilitation; metabolic rate; sport
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation intervention group (Active Comparator): The group is performing a strength endurance training intervention in addition with rehabilitation exercise intervention.
  Interventions: Other: rehabilitation exercise intervention
- Placebo rehabilitation (Placebo Comparator): The group is performing a strength endurance training intervention in addition with placebo rehabilitation exercise intervention.
  Interventions: Other: placebo control group

INTERVENTIONS:
Other: rehabilitation exercise intervention — exercise intervention: 15 minutes warm up, 30 minutes strength endurance training, 60 minutes rehabilitation exercise training - once a week
  15 minutes warm up, 30 minutes strength endurance training - once a week
  Arms: Rehabilitation intervention group
Other: placebo control group — exercise intervention: 15 minutes warm up, 30 minutes strength endurance training, 5 minutes walking 55 minutes conversation in the group- once a week
  15 minutes warm up, 30 minutes strength endurance training - once a week
  Arms: Placebo rehabilitation

SUMMARY:
The purposes of the study are

* to determine if a supervised exercise intervention is improving the metabolic parameters in type 2 diabetes patients
* to investigate what kind of intervention (strength endurance training versus combined strength endurance training and rehabilitation exercise intervention)is more effective in improving the metabolic parameters in patients with type 2 diabetes
* to assess which exercise intervention induces higher effects to the metabolic rate and cardiac and pulmonary capacity
* to investigate what kind of intervention includes highest effects in long term persistence of these positive effects

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes (ADA criteria)
* admitted diabetes treatment will be diet and oral hypoglycemic agents

Exclusion Criteria:

* sports intervention > 60 minutes per week

medical conditions

* proliferative retinopathy
* instable coronary heart disease
* acute clinically significant intercurrent disease
* inability to perform scheduled physical activity programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
alteration of HbA1c-level (haemoglobin A1c) | 6 months

SECONDARY OUTCOMES:
alteration of total cholesterol level | 6 months
alteration of LDL-cholesterol-level | 6 months
alteration of HDL-cholesterol-level | 6 months
alteration of triglyceride-level | 6 months
alteration of antidiabetic medications | 6 months
alteration of anthropometry | 6 months
  body weight; body mass index; hip-to-waist-ratio
alteration of body composition | 6 months
  measured by Bio-impedance analysis
alteration of resting metabolic rate | 6 months
  1. measured by Spirometrie (Cortex metamax)
  2. calculated by Bio-impedance analysis (TANITA)
alteration of blood pressure | 6 months
alteration of cardiac and pulmonary capacity | 6 months
  1. measured by ergometry
  2. six-minutes walk test
alteration of quality of life | 6 months
follow up of all parameters mentioned above | 15 months
  follow up after 15 months without any supervised intervention

CONTACTS AND LOCATIONS:
Overall Officials: Andree Hillebrecht, Dr. med., Study Chair — University of Giessen; Dusan Hamar, Prof. Dr., Study Director — Comenius University
Locations (2):
- Germany (2):
  - University of Giessen, Giessen, Hesse
  - Sportpark Zwickau, Glauchau, Meerane, Zwickau, Saxony